CLINICAL TRIAL: NCT01287663
Title: Effectiveness of Permethrin Impregnated Underwear in Preventing Louse Proliferation in Infected Homeless
Acronym: ERPOUPER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-A01406-33; 2010 30 (Other: AP HM)
Record Dates: First submitted 2011-01-31; First posted 2011-02-01 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Body's Louses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- no permethrin (Placebo Comparator)
  Interventions: Drug: no Permethrin impregnated
- permethrin (Experimental)
  Interventions: Drug: Permethrin impregnated

INTERVENTIONS:
Drug: Permethrin impregnated
  Arms: permethrin
Drug: no Permethrin impregnated
  Arms: no permethrin

SUMMARY:
Homelessness, also name the fourth world, is a growing public health problem worldwide. Previous studies showed that up to 30% of the homeless people reported pruritus that often results in itchy lesions, which expose them to bacterial skin infections.

The investigators therefore conducted a randomized, double-blind, placebo-controlled trial to test the hypothesis that a single oral dose of ivermectin was effective in significantly reducing the prevalence of pruritus in a sheltered homeless population.

ELIGIBILITY:
Inclusion Criteria:

* Patient HOMELESS PERSON " individual who has no regular access to a conventional residence ", appearing during the period of study at reception centers (Forbin or Madrague Ville) and being in the habit of wearing there (at least 4 times a week),
* Male genital organ and feminine,
* Of more than 18 years old,
* Presenting of the prurit, hurts of scratching or the louses
* Wishing to change his underwear,
* Having given his lit(enlightened) consent

Exclusion Criteria:

* Woman presenting a sexually transmitted infection (infection with gonococcus, with Chlamydia trachomatis, with Trichomonas vaginalis) revealing on the takings realized during the consultation of inclusion but the bacteriological results of which will be known only secondarily.
* Pregnant Woman presenting to the consultation of inclusion of métrorragies either a break of the pocket of waters or an infectious complication of the pregnancy.
* Woman removing her consent during the study.
* Lost sight Woman.
* Woman deprived of freedom, judicial or administrative;
* Woman hospitalized for quite other reason that looks for her(it);
* Woman hospitalized in a sanitary establishment or social in the other purposes that the research;
* Major Woman except state to express its consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Show that underwear soaked with permethrine in 8 % allow to reduce in a long-lasting way (J90 and J365) of 50 % the index of infestation and prevalency of the louses in the group treated with regard to the group placebo. | 2 YEARS

SECONDARY OUTCOMES:
Show that underwear soaked with permethrine in 8 % allow to reduce in a long-lasting way (J90 and J365) of 50 % the index of infestation and prevalency of the louses in the group treated with regard to the group placebo. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Benkouiten S, Drali R, Badiaga S, Veracx A, Giorgi R, Raoult D, Brouqui P. Effect of permethrin-impregnated underwear on body lice in sheltered homeless persons: a randomized controlled trial. JAMA Dermatol. 2014 Mar;150(3):273-9. doi: 10.1001/jamadermatol.2013.6398. PMID 24305799